CLINICAL TRIAL: NCT05960084
Title: Impact of Reducing Colistin Use on Colistin Resistance in Humans and Poultry in Indonesia
Acronym: COINCIDE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Indonesia University (Other); Center For Indonesian Veterinary Analytical Studies (Unknown); Utrecht University (Other); Institute of Tropical Medicine (Other Government); University of Calgary (Other); Directorate of Veterinary Public Health, Ministry of Agriculture (Unknown)
Responsible Party: Principal Investigator, Juliëtte Severin, Associate professor, Medical coordinator Unit infection prevention, Erasmus Medical Center
Other Study IDs: 22-03-0255
Record Dates: First submitted 2023-06-16; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Colonization, Asymptomatic; Colistin; Mcr-1; Antimicrobial Resistance
Keywords: Escherichia coli
MeSH Terms: conditions — Asymptomatic Infections; Escherichia coli Infections | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bacterial DNA, particularly E. coli
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: screening — screening for colistin resistant E. coli

SUMMARY:
Colistin (polymyxin E) is considered a last resort antimicrobial for treatment of infections with multidrug- resistant bacteria, classified by WHO as 'highest prioritized, critically important for human medicine'. WHO suggests to ban or highly restrict its use in animals. In Indonesia, colistin resistance in human Escherichia coli isolates is poorly characterized as it requires specific non-routine tests. Presence of colistin resistance in E. coli in poultry resulted in a ban for livestock in Indonesia in 2020. However, colistin is still suspected to be routinely used in humans in multiple settings but the reasons for these practices are poorly understood. The ban on colistin use in livestock offers a unique opportunity to assess the impact of this intervention on colistin resistance in humans and animals, and how a One Health perspective can strengthen this intervention. This project aims to: i) determine phenotypic and genotypic colistin resistance in E. coli from humans and poultry in Indonesia; ii) assess the impact of the colistin ban on resistance in E. coli in animals and humans; iii) estimate the transmission of colistin resistance between animals and humans; iv) study colistin use and perceptions at the community level; and v) expand the initial colistin ban in the animal production sector into an integrative multi-sectorial One Health intervention, which will be designed and implemented using a community participatory approach. This project will provide a strong scientific basis to AMR policies in Indonesia, with great significance across Southeast Asia.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with age >= 18 years old, that are willing to participate

Exclusion Criteria:

* Vomiting and/or diarrhea

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Local public health centers (Puskesmas) will be recruiting participants and sampling in the three districts of Central Java in Indonesia: Sukoharjo, Klaten, and Karanganyar. The targeted study participants are individuals at least 18 years old without any diarrhea and/or vomiting at the time of visit to local public health centers. In addition, poultry farms will be approached for sampling in the same area.
Sampling Method: Non-Probability Sample
Enrollment: 803 (Estimated)
Dates: Start 2023-07-23 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mcr-positive E. coli in humans in the community in Central Java, Indonesia | 2024
  Carriage of mcr-1 positive E. coli will be measured by taking rectal swabs of participants for bacterial culture.
Risk factors associated with carriage of mcr-positive E. coli in humans | 2024
  Interviews based on structured close-ended questionnaires will be used. The questionnaire will include demographic data (gender, age) and possible risk factors (underlying diseases, certain habits as smoking, job, previous antibiotic use).

SECONDARY OUTCOMES:
Transmission of mcr-positive E. coli between farmers and poultry | 2024
  Transmission will be investigated by analyzing the mcr-positive E. coli with genomic analysis, such as whole genome sequencing.
Overall antibiotic prescription behaviour in public health centers in Central Java, Indonesia | 2024
  Several methods will be used, including the drug-bag method, and collection of antibiotic prescription per public health center.

CONTACTS AND LOCATIONS:
Overall Officials: Anis Karuniawati, MD PhD, Principal Investigator — Indonesia University
Locations (1):
- Faculty of Medicine, University of Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The study will be carried our according to the principles states in the Declaration of Helsinki (Ethical Principles for Medical Research Involving Human Subjects), all applicable regulations and according to established international and national scientific standards.